CLINICAL TRIAL: NCT06256328
Title: A Randomized, Multicenter, Double-blind, Phase II Study to Compare the Efficacy and Safety of the Treatment With ONO-4578 in Combination With Nivolumab, Fluoropyrimidine-based and Platinum- Based Chemotherapy (Hereinafter Referred to as Chemotherapy) With Those of the Treatment With Placebo in Combination With Nivolumab and Chemotherapy in Chemotherapy-naïve Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Unresectable Advanced or Recurrent Gastric Cancer (Including Esophagogastric Junction Cancer)
Brief Title: A Study to Investigate the Efficacy and Safety of ONO-4578 in Combination With Nivolumab and Chemotherapy in Chemotherapy-naïve Participants With HER2-negative Unresectable Advanced or Recurrent Gastric Cancer (Including Esophagogastric Junction Cancer)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONO-4578-08
Record Dates: First submitted 2024-01-23; First posted 2024-02-13 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine; S 1 (combination); Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ONO-4578+Nivolumab+chemotherapy (Experimental)
  Interventions: Drug: ONO-4578; Drug: Oxaliplatin; Drug: Capecitabine; Drug: S-1; Drug: Nivolumab
- placebo+Nivolumab+chemotherapy (Placebo Comparator)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: S-1; Drug: Nivolumab; Drug: Placebo

INTERVENTIONS:
Drug: ONO-4578 — Specified dose, once daily
  Arms: ONO-4578+Nivolumab+chemotherapy
Drug: Oxaliplatin — Specified dose on specified days
Drug: Capecitabine — Specified dose on specified days
Drug: S-1 — Specified dose on specified days
  Other Names: Tegafur-gimeracil-oteracil potassium
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
Drug: Placebo — Specified dose, once daily
  Arms: placebo+Nivolumab+chemotherapy

SUMMARY:
This study is to compare and evaluate the efficacy and safety of the treatment with ONO-4578 in combination with nivolumab and chemotherapy with those of the treatment with placebo in combination with nivolumab and chemotherapy in chemotherapy-naïve participants with HER2- negative unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer).

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric or esophagogastric junction cancer histologically diagnosed as adenocarcinoma
* Patients have not been treated with systemic chemotherapy as first-line therapy
* Patients who can provide tumor tissue samples

Exclusion Criteria:

* Patients unable to take oral medicines
* Patients with HER2-positive
* Patients with contraindications to nivolumab, oxaliplatin, S-1, or capecitabine
* Patients who have a history of severe drug-related adverse reactions caused by non- steroidal anti-inflammatory drugs (NSAIDs) or who have complications caused by NSAIDs requiring treatment
* Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease, such as rheumatoid arthritis
* Patients with headache and/or nausea associated with brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (site investigator assessment) | up to 2years

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2years
Objective response rate (ORR) (site investigator assessment) | up to 2years
Best overall response (BOR) (site investigator assessment) | up to 2years
Duration of response (DOR) (site investigator assessment) | up to 2years
Disease control rate (DCR) (site investigator assessment) | up to 2years
Time to response (TTR) (site investigator assessment) | up to 2years
Maximum percent change in the sum diameters of the target lesions (site investigator assessment) | up to 2years
Progression-free survival after the next line of therapy (PFS2) (site investigator assessment) | up to 2years
Adverse event (AE) | Up to 30 days after the last dose
  Number of participants with treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (63):
- Japan (32):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - NHO Kyushu Cancer Center, Fukuoka, Fukuoka
  - JCHO Kyushu Hospital, Yahatanishi-ku, Kitakyusyu-shi, Fukuoka
  - Gunma Prefectural Cancer Center, Ota-shi, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - JOHAS Kansai Rosai Hospital, Amagasaki-shi, Hyōgo
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital, Kasama-shi, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Yahaba-cho, Shiwa-gun, Iwate
  - Kagawa University Hospital, Miki-cho, Kita-gun, Kagawa-ken
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaki Citizen Hospital, Osaki-shi, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Osaka International Cancer Institute, Chuo-ku, Osaka
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Kindai University Hospital, Sayama-shi, Osaka
  - Osaka General Medical Center, Sumiyoshi-ku, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Saitama Cancer Center, Ina-machi, Kitaadati-gun, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Sunto-gun, Shizuoka
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - IMSUT Hospital, The Institute of Medical Science, The University of Tokyo, Minato-Ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Osaka Metropolitan University Hospital, Osaka
- South Korea (25):
  - Kosin University Gospel Hospital, Busan, Gangwon-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeonbuk national university hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No